CLINICAL TRIAL: NCT06644313
Title: Vebreltinib for Neoadjuvant in MET-altered Stage IIIA-IIIB (N2) Non-small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of thoracic department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-025
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Potentially Resectable MET-altered Non-Small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer Stage III; Non-small Cell Lung Cancer with MET mutation; Neoadjuvant; Vebreltinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: All enrolled patients received Vebreltinib neoadjuvant therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vebreltinib (Experimental)
  Interventions: Drug: Vebreltinib

INTERVENTIONS:
Drug: Vebreltinib — Neoadjuvant treatment stage: Vebreltinib 200mg, bid, po, 2-4 months in total; Surgical treatment stage: CR + PR patients and SD + PD patients who could still undergo surgery will receive radical surgery; Adjuvant treatment stage: CR, PR and SD patients who have been treated surgically: Vebreltinib 200mg, bid, po, up to 2 years/until the disease progressed. PD patients: transferred into medical oncology or/and radiation oncology and receive comprehensive therapy.

SUMMARY:
According to the 2024 edition of the NCCN guidelines and the 2023 edition of the CSCO guidelines, perioperative treatment is recommended for patients with stage IIIA and IIIB (T3N2) non-small cell lung cancer (NSCLC). Targeted therapies for NSCLC, such as EGFR inhibitors and ALK inhibitors, have been explored in the neoadjuvant setting. For patients with MET alterations, some have undergone preoperative MET inhibitor treatment, achieving pathological downstaging followed by surgery, resulting in R0 resection. Therefore, this is a prospective, cohort, single-center phase II clinical study to evaluate the efficacy and safety of Vebreltinib as a neoadjuvant treatment for patients with MET-altered stage IIIA-IIIB (N2) NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient shall sign the Informed Consent Form. 2.Aged 18 ≥ years. 3.Histological or cytological diagnosis of NSCLC by needle biopsy, and evaluated by researchers as stage III-IVA.

  4.NGS gene testing confirmed MET alterations, which include the following two types: Cohort 1: MET exon 14 skipping mutations (NGS results from tissue or blood samples certified by CLIA or CAP-approved laboratories); Cohort 2: Primary MET amplification (NGS results or FISH results from tissue or blood samples certified by CLIA or CAP-approved laboratories)..

  5.Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1. 6. According to the MDT evaluation (which should include a thoracic surgeon specializing in tumor surgery), it is considered that the primary NSCLC is potentially completely resectable; 7. At least 1 measurable lesion according to RECIST 1.1. 8.Patients with good function of other main organs (liver, kidney, blood system, etc.) 9.Patients with lung function can tolerate surgery; 10.Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative. 11. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 d

Exclusion Criteria:

* 1. Previously received targeted therapy (including TKI or monoclonal antibodies), immunotherapy, or any investigational drug treatment for NSCLC; 2.Pathological confirmation of mixed small cell and non-small cell lung cancer; 3.Patients with a malignancy other than NSCLC within five years prior to the start of this trial，except for cured basal cell carcinoma of the skin, early gastrointestinal (GI) carcinoma excised through endoscopy, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary thyroid carcinoma, or any cured cancer deemed to have no impact on the survival of the current NSCLC; 4.Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases; 5.Patients with congenital or acquired immune dysfunction (such as HIV infected individuals); 6.Received other major surgical treatments (excluding diagnosis) within 4 weeks prior to the start of the study or expected to undergo major surgical treatments during the study period; 7.Participants who are allergic to the test drug or any auxiliary materials; 8.A history of extensive diffuse bilateral interstitial fibrosis in the past or before medication, or a known grade 3 or 4 history of interstitial fibrosis or interstitial lung disease, including pneumonia, allergic pneumonia, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not including local radiation pneumonia or radiation pulmonary fibrosis history;8. Pregnant or lactating women; 9.Any malabsorption; 10.Participants suffering from nervous system diseases or mental diseases that cannot cooperate 11.Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response (ORR) rate | up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 30 months
  DCR Rate is defined as the proportion of patients who achieve stable disease (SD), partial response (PR), or complete response (CR) among all patients.
Major pathologic response (MPR) rate | Up to 30 months
  MPR rate is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants.
Pathologic complete response (PCR) rate | Up to 30 months
  PCR rate is defined as the proportion of participants who have achieved pathologic complete response (on routine hematoxylin and eosin staining, no tumor cell can be found in tumor bed or lymph node) in all participants.
Event-free survival (EFS) | up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
3-year overall survival (OS) | Up to 36 months
  OS is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Overall survival (OS) | up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.

OTHER OUTCOMES:
The correlation between stratification factors such as disease stage, smoking history, and treatment efficacy | Up to 30 months
  The correlation between stratification factors such as disease stage, smoking history, and treatment efficacy.

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.